CLINICAL TRIAL: NCT06052696
Title: Adjuvant Nonavalent HPV Vaccination in Women Treated for Vulvar HSIL, a Randomised Placebo Controlled Trial
Brief Title: Adjuvant Nonavalent HPV Vaccination in Women Treated for Vulvar HSIL
Acronym: VulVaccin
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Ralf van de Laar, MD, gynaecologic oncologist., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MEC-2023-0526; 2023-506792-94-00 (Other: EMA)
Record Dates: First submitted 2023-08-31; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Vulvar HSIL; HPV
Keywords: HPV; VHSIL; Vaccination
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gardasil 9 (Experimental): see intervention
  Interventions: Drug: Gardasil 9 Suspension for Injection
- placebo (Placebo Comparator): see intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gardasil 9 Suspension for Injection — After randomisation in the Gardasil arm, women will receive 3 Gardasil vaccinations
  1. First injection: preferable at time of start treatment (imiquimod, lase or surgery). Window 4 weeks prior to treatment start (because surgical treatment can be postponed for logistical reasons) and 4 weeks after start treatment.
  2. Second injection: should be administered at least 1 month after the first injection and 3 months before the third injection.
  3. Third injection should be administered at 3 months after second injection. All injections should be administered within 1 year.
  Arms: Gardasil 9
Drug: Placebo — After randomisation in the PLacebo arm, women will receive 3 Placebo vaccination with NaCl 0.9%
  1. First injection: preferable at time of start treatment (imiquimod, lase or surgery). Window 4 weeks prior to treatment start (because surgical treatment can be postponed for logistical reasons) and 4 weeks after start treatment.
  2. Second injection: should be administered at least 1 month after the first injection and 3 months before the third injection.
  3. Third injection should be administered at 3 months after second injection. All injections should be administered within 1 year.
  Arms: placebo

SUMMARY:
Problem description:

Yearly, approximately 45000 women develop vulvar cancer worldwide. It is estimated that about 30% of all vulvar carcinomas are HPV related. As with other HPV related (pre)malignancies, the incidence has been rising over the past 20 years. The peak incidence of premalignant lesions of the vulva, also called Vulvar High Grade Squamous Intraepithelial Lesion (vHSIL), lies between 35 and 40 years of age. Multiple treatments are available, including surgery, laser vaporization, and topical imiquimod, with comparable success rate. Despite treatment, at least 30% of women will develop a recurrence within 2 years, with a much higher lifetime risk of recurrence. This results in multiple treatments with sometimes disfiguring effects and associated negative psychosocial and psychosexual impact. Woman with vulvar HSIL have a lifelong increased risk of vulvar cancer, and approximately 10% of women with (treated) vulvar HSIL will develop vulvar cancer within 10 years of first diagnosis. The risk of malignancy is significantly higher in women with recurrent disease, compared to women without recurrence.

Solution / research direction, To date, a successful strategy for reduction of recurrences of HSIL has not been established. The available positive evidence on the use of concurrent HPV vaccination in the treatment of vulvar HSIL is rising, yet insufficient to guide clinical practice. There is limited data that prophylactic HPV vaccination after treatment of vulvar HSIL reduces the chance of recurrence, therefore leading to a reduction in repeated (surgical) interventions. There are no randomised controlled studies supporting this data.

Aim The aim of current project is to determine the effectiveness of nonavalent HPV vaccination versus placebo in preventing recurrence in women treated for vulvar HSIL.

Plan of investigation This is a randomised, double blinded, placebo controlled trial in women treated for vulvar HSIL. Adult female patients, diagnosed with vulvar HSIL planned for treatment and no prior HPV vaccination will be included. Randomisation will be in a 1:1 ratio to additional nonavalent HPV vaccination versus additional placebo vaccination.

Expected outcome. Based on previous non-randomised studies, a significant reduction in recurrences, improvement of quality of life and a reduction of economic burden of the disease is expected.

ELIGIBILITY:
Inclusion criteria

* Women 18 years or older
* Vulvar High-grade Squamous Intraepithelial Lesion (vHSIL), histologically proven
* Planned for treatment (surgical, laser or imiquimod) for vHSIL

Exclusion criteria

* Prior HPV vaccination
* (Micro-) invasive carcinoma or history of HPV related genital carcinoma (cervix, anal, vulva)
* Pregnancy
* Women allergic to vaccine components
* HIV infection
* Immune compromised patients (currently on immunosuppressive medication

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Does additional HPV vaccination reduce the recurrence of vHSIL compared to placebo? | 24 months after last inclusion
  Difference in number and percentage of patients with clinical recurrence rate of vulvar HSIL between HPV vaccination and placebo at 6 and 12 months

SECONDARY OUTCOMES:
1. What is the effectiveness (complete remission) after treatment in vaccination versus placebo at 6 and 12 months? | 6 and 12 months after last inclusion
  1. Difference in number and percentage of patients with clinical recurrence rate of vulvar HSIL between HPV vaccination and placebo at 6 and 12 months
2. What is the effectiveness (complete remission) after treatment in vaccination versus placebo at 6 and 12 months in primary episode vHSIL versus recurrence? | 6 and 12 months after last inclusion
  2. Difference in number and percentage of patients with clinical recurrence rate of vulvar HSIL between HPV vaccination and placebo at 6 and 12 months for primary vHSIL versus recurrent vHSIL.
3. What is the effectiveness of adjuvant vaccination in different treatments of vHSIL (laser, imiquimod, excision) at 24 months? | 24 months after last inclusion
  3. Difference in number and percentage of patients with clinical recurrence rate of vulvar HSIL between the different treatment modalities
4. How often is additional treatment for vHSIL needed in the study period? Is this different between the study groups? | 24 months after last inclusion
  4. Difference in number and percentage for additional treatment necessary after primary treatment.
5. What is the effect of vaccination versus placebo on different HPV types (HPV type of primary and recurrence)? | 24 months after last inclusion
  5. Description and percentage of different HPV types. Percentage clearance of primary HPV type for vaccination versus placebo.
6. What is the level of antibodies at baseline and after (placebo) vaccination? | 24 months after last inclusion
  6. Number of antibodies and percentage of increase or decrease after vaccination compared to antibodies before vaccination. Is there correlation between number or percentage of recurrence. Is that different in primary versus recurrent episode vHSIL
7. Is the intervention cost effective? | 24 months after last inclusion
  7. incremental cost-effectiveness ratio (ICER), described the difference in costs and budget impact analysis
8. Is Quality of life (measured with Euroqol 5D-5L questionnaire) improved after vaccination compared to placebo? | 24 months after last inclusion
  8.Description and change in numeric value and percentage in different score form questionnaires. Percentage increase of decrease QoL
8. Is sexual health (measured with Female Sexual Function Index, FSFI questionnaire) improved after vaccination compared to placebo? | 24 months after last inclusion
  8.Description and change in numeric value and percentage in different score form questionnaires. Percentage increase of decrease sexual impact
9. What is the effect of vaccination versus placebo on CIN/cervical cytology of the uterine cervix? | 24 months after last inclusion
  9. Difference number and percentage in HPV types cervical cytology and vHSIL before and after vaccination.
10. Long-term follow-up: Is there a difference between vaccination and placebo group in number of recurrences of vHSIL (5 and 10 years) and the occurrence of vulvar malignancies (2, 5 and 10 years)? | 5 and 10 year
  10. Difference in number and percentage in recurrence rate of vulvar HSIL and vulvar cancer between HPV vaccination and placebo. Other HPV related disease known?

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vaessen VJGM, van de Laar RLO, Piso-Jozwiak M, Dalm VASH, Joura EA, Jentschke M, van Beekhuizen HJ. Adjuvant nonavalent HPV vaccination in women treated for vulvar HSIL, a randomized placebo-controlled trial; VulVaccin study protocol. BMC Cancer. 2025 May 20;25(1):903. doi: 10.1186/s12885-025-14275-w. PMID 40394508